CLINICAL TRIAL: NCT04323774
Title: AYA-RISE: Refining a Scalable, Patient- and Family-centered Intervention to Improve Cancer Risk Communication and Decision-making Among Adolescents and Young Adults With Cancer Risk Syndromes
Brief Title: Intervention For AYAS With Cancer Risk Syndromes
Acronym: AYA-RISE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Mack, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-003; U01CA243688-01 (NIH)
Record Dates: First submitted 2020-03-23; First posted 2020-03-27 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Cancer Risk Syndrome
Keywords: Cancer Risk Syndrome; LiFraumeni Syndrome Association (LFSA) Youth Conference
MeSH Terms: interventions — Genetic Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Aim 1-Part 1 Stakeholder Interview (No Intervention): This arm will focus on finding the best format for the study intervention (called AYA-RISE) whether AYA-RISE is easy to use; and whether patients, family caregivers, and providers find AYA-RISE acceptable.
  The research study procedures include:
  * Using and reviewing AYA-RISE
  * Participating in audio-recorded, 30-minute interviews
- Aim 1-Part 2 (Experimental): This arm is a pilot study of the study intervention (called AYA-RISE).
  The activities involved in this part of the study are:
  * Baseline Questionnaire
  * Using and reviewing AYA-RISE
  * Follow-up Questionnaire
  * Brief interviews to get feedback on AYA-RISE
  Interventions: Behavioral: AYA-RISE Adolescents and Young Adults Risk Information and Screening Education
- Aim 2-Genetic Counseling (Active Comparator): The names of the study activities involved in this study are:
  * Baseline Questionnaire
  * Follow-up Questionnaire
  * Medical record review
  The study procedures will all take place on the day of the patient's regularly scheduled clinic visit. Participants will be in this research study for up to 1 year.
  Interventions: Behavioral: Standard clinical visit for genetic counseling
- Aim 2- Genetic Counseling with AYA-RISE (Experimental): The names of the study activities involved in this study are:
  * Baseline Questionnaire
  * Follow-up Questionnaire
  * Medical record review
  * Using the study intervention, AYA-RISE
  The study procedures will all take place on the day of the patient's regularly scheduled clinic visit. Participants will be in this research study for up to 1 year.
  Interventions: Behavioral: AYA-RISE Adolescents and Young Adults Risk Information and Screening Education
- Aim 3 Semi-structured interviews (No Intervention): Each site will conduct 30-minute interviews with patients, caregivers, and providers, and site principal investigators.

INTERVENTIONS:
Behavioral: AYA-RISE Adolescents and Young Adults Risk Information and Screening Education — A chatbot is a computer program that can chat with humans. The text the chatbot uses to talk with humans was created by real people, but the chatbot itself is not a real person. A company called Clear Genetics developed the original chatbot and patient portal, and this study team customized it for this research study.
  Other Names: AYA-RISE
  Arms: Aim 1-Part 2; Aim 2- Genetic Counseling with AYA-RISE
Behavioral: Standard clinical visit for genetic counseling — Standard clinical visit for genetic counseling and follow up
  Arms: Aim 2-Genetic Counseling

SUMMARY:
This research is being done because there is a need to improve cancer risk communication and decision-making among adolescents and young adults. In this study, the investigators are looking at whether using a chatbot and online portal for cancer risk information helps improve communication and decision-making.

* Over 70,000 adolescents and young adults (AYAs) are diagnosed with cancer in the U.S. every year and up to 10% have genetic changes (or, mutations) that put them at a higher risk of developing new cancers during their lifetimes. These genetic mutations can result in cancer risk syndromes (such as, Lynch Syndrome or Li-Fraumeni Syndrome). Identifying cancer risk syndromes can allow for screening and early diagnosis of future cancers, which could ultimately save lives and offer more care choices for patients. As a result, genetic counseling and testing for cancer risk syndromes is being recommended more for Adolescents and Young Adults with new cancer diagnoses, regardless of family history.
* This research study to develop an intervention called AYA-RISE that aims to assist AYAs with cancer risk communication and decision-making around their caregivers.

DETAILED DESCRIPTION:
This research study involves three aims (Aims 1, 2, and 3).

* Aim 1, Part 1, which focuses on finding the best format for the study intervention (called AYA-RISE); whether AYA-RISE is easy to use; and whether patients, family caregivers, and providers find AYA-RISE acceptable.The research study procedures include:

  * Using and reviewing AYA-RISE,
  * Participating in audio-recorded, 30-minute interviews
* Aim 1, Part 2, which is a pilot study of the study intervention (called AYA-RISE). In this pilot study, the investigators are looking at whether AYA-RISE is easy to use and what participants think of it.

  -- The activities involved in this part of the study are:
  * Baseline Questionnaire
  * Using and reviewing AYA-RISE
  * Follow-up Questionnaire
  * Brief feedback interviews on AYA-RISE
* In Aim 2, participants will be randomized trial into one of two groups;

  * Group 1: Standard Genetic Counseling/follow-up visit or
  * Group 2 : Standard Genetic Counseling/follow-up visit and Access to AYA-Rise
* Aim 3: Semi-Structured Interviews:

  * Evaluate implementation outcomes using 28 semi-structured interviews with patients, family members, providers, and site principal investigators

ELIGIBILITY:
Inclusion Criteria:

* Across all study aims, we will enroll AYA patients, family members/caregivers, and providers.

AIM 1, PART 1 - STAKEHOLDER INTERVIEWS

AYA Patients

1. Ages 12-24 years, inclusive
2. Diagnosed with a cancer risk syndrome
3. English-speaking and -reading
4. Receiving care at any of the study sites OR participating in the LiFraumeni Syndrome Association (LFSA) Youth Conference
5. Adequate cognitive function per NeuroQOL indicated by a score of 30 or greater
6. Not receiving active cancer therapy

Family caregivers-Inclusion Criteria

1. Parent/guardian, spouse/partner, or other family member who participates in the care of AYAs aged 12-24 with cancer risk syndromes
2. English-speaking and -reading
3. At any of the study sites

Providers Inclusion Criteria (Oncologists, nurses, genetic counselors, social workers, or psychologists)

1. English-speaking and reading
2. Caring for AYAs aged 12-24 with cancer risk syndromes at any of the study sites

AIM 1, PART 2 - INTERVENTION PILOT

AYA Patients

1. Ages 12-24 years, inclusive
2. Diagnosed with a cancer risk syndrome
3. English-speaking and -reading
4. Receiving care at Dana-Farber Cancer Institute
5. Adequate cognitive function per NeuroQOL, indicated by a score of 30 or greater
6. Not receiving active cancer therapy
7. Did not participate in a stakeholder interview

Eligibility notes:

* Family caregivers of participating 12-17y patients will be eligible to participate in the pilot
* 12-17y patients can participate without a family member if both the patient and family member agree.
* Patients 18-24y will have the option to participate with or without a family member.

AIM 2 - RANDOMIZED TRIAL

AYA Patients

1. Ages 12-24 years, inclusive
2. Diagnosed with a cancer risk syndrome
3. English-speaking and reading
4. Has a planned post-disclosure genetic counseling or follow-up visit at any of the study sites
5. Adequate cognitive function per NeuroQOL, indicated by a score of 30 or greater
6. Not receiving active cancer therapy
7. Did not participate in either part of Aim 1 (interview or pilot)

Family caregivers

1. Parent/guardian, spouse/partner, or other family member who participates in the care of AYAs aged 12-24 with cancer risk syndromes
2. English-speaking and -reading
3. At any of the study sites
4. Did not participate in either part of Aim 1 (interview or pilot)

AIM 3 - SEMI-STRUCTURED INTERVIEWS AYA Patients, Family Caregivers, Providers, and Site PIs

1. Participated in the intervention arm of Aim 2, or
2. Is a site principal investigator at one of the 4 participating study sites

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Consenting AYA use AYA-RISE | 2 years
  The feasibility (>70% consenting AYAs use AYA-RISE through the risk communication step of the chat and patient portal, based on use data from Clear Genetics)
Percentage of Acceptability | 2 years
  Acceptability (>70% AYAs consider the intervention acceptable, measured as a post-test AIM score >4.)
Change in patient knowledge of cancer risk and screening | baseline to post-visit surveys up to 24 months
  This change will be measured by baseline and post-visit survey responses on the Knowledge of Cancer Screening and Gist Comprehension of Genetic Cancer Risk measures.
Change in psychological distress | baseline to post-visit surveys up to 24 months
  This change will be measured by baseline and post-visit survey responses using the psychosocial aspects of hereditary cancer (PAHC) measure.
Patient ownership of information in the intervention arm | 24 Months
  determined as % AYAs able to store and access portal information
Participants who followed up for recommended care | screening and follow-up over the next year up to 24 Months
  We will identify recommended care and screening via medical record review, and whether care was received, post-visit.
Utilization of AYA-RISE | 2 Years
  Chat transcripts and patient portal access
Acceptability of AYA-RISE | 2 Years
  Semi-structured interview: How did patients, providers, family members feel about the intervention? Was the experience positive, negative, or neutral? An analytic matrix on intervention design will be used to code of semi-structured interviews
Adoption of AYA-RISE | 2 Years
  An analytic matrix on intervention design will be used to code of semi-structured interviews
  - Semi-structured interview of Providers and Clinic Leaders
  * Were patients and providers willing to try the intervention?
  * Would they want to continue to use the intervention?
Practicality of Using AYA-RISE | 2 Years
  An analytic matrix on intervention design will be used to code of semi-structured interviews: Site PI Semi-structured interview
  * Is it practical to continue to use AYA-RISE within constraints of
  * clinic, provider, and patient/family needs?
Fidelity of AYA-RISE | 2 Years
  * Site RA: Observation and Checklist
  * Does actual implementation match the planned process?
Sustainability of AYA-Rise | 2 Years
  An analytic matrix on intervention design will be used to code of semi-structured interviews Can the processes required for AYA-RISE be maintained beyond the research setting?

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mack, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu